CLINICAL TRIAL: NCT06029894
Title: Improving Sleep and Alzheimer's Disease (AD) Biomarkers: A Pilot Randomized Clinical Trial (RCT) of Citicoline
Brief Title: Improving Sleep and AD Biomarkers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Victoria Pak, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00006047; 1R61AG080606-01 (NIH)
Record Dates: First submitted 2023-08-10; First posted 2023-09-08 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Dementia; Citicoline supplement
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Citicoline and placebo treatment will be blinded. The study treatment will be labeled using a unique Kit ID number that is linked to a randomization scheme. The active and placebo tablets will be identical and presented in the same packaging to ensure the blinding of the study medication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants with MCI will receive dietary citicoline supplements.
  Interventions: Dietary Supplement: Citicoline Supplement
- Placebo (Placebo Comparator): Participants with MCI will receive a placebo supplement.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Citicoline Supplement — Participants with MCI will receive dietary citicoline supplements. Subjective sleep measures will be measured via the Pittsburgh Sleep Quality Index (for measurement of sleep quality) and Epworth Sleepiness Scale (for measurement of sleepiness). Cognition will be measured by Rey Auditory Verbal Learning Test (RAVLT), Trail Making Test (TMT) Parts A & B, and the Montreal Cognitive Assessment (MOCA). Participants will complete all questionnaires at baseline and at follow-up at 3 months. Participants will undergo a blood draw of approximately 20 ml at baseline and at follow-up.
  Other Names: Citicoline 1000mg
  Arms: Treatment Group
Other: Placebo — Participants with MCI will receive a placebo supplement. Subjective sleep measures will be measured via the Pittsburgh Sleep Quality Index (for measurement of sleep quality) and Epworth Sleepiness Scale (for measurement of sleepiness). Cognition will be measured by Rey Auditory Verbal Learning Test (RAVLT), Trail Making Test (TMT) Parts A & B, and the Montreal Cognitive Assessment (MOCA). Participants will complete all questionnaires at baseline and at follow-up at 3 months. Participants will undergo a blood draw of approximately 20 ml at baseline and at follow-up.
  Arms: Placebo

SUMMARY:
The purpose of this research is to learn whether a dietary citicoline supplement will impact sleep and cognition. Cognitive disorders include such things as memory disorders and mild cognitive impairment. The investigators are studying persons with mild cognitive impairment (MCI). For this population, the team will assess whether citicoline also impacts biomarkers, a marker of the patient's biological state, in their body.

The investigators are interested in learning more about a dietary supplement called citicoline and how it helps sleep, cognition, and markers of Alzheimer's. Previous studies have evaluated this dietary supplement and shown that citicoline may impact cognitive decline. The investigator would like to evaluate if citicoline will also impact sleep and markers of Alzheimer's. This dietary supplement has been assessed in older adults and found to be well tolerated. Citicoline has been used safely in cognitive impairment populations at the same dosage.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled pilot trial. To assess the hypothesis in this proposed study, the investigator will leverage infrastructure from the Emory Alzheimer's disease research center (ADRC), ADRC-affiliated centers, mild cognitive impairment, related research cohorts with potential eligible participants interested in participating in future studies, the Emory Sleep Center, and also recruit from the community. The research team will be actively recruiting individuals with MCI with confirmed medical diagnoses. The investigator will also collect data from personal interviews on prior medical diagnoses from the medical record along with current medication usage. Researchers will also obtain available baseline AD biomarker data from participants at baseline if they have cerebrospinal fluid (CSF) and/or blood data available on AD biomarkers within the past year from prior research studies, the investigators will use this data for the study records which will serve as their 'baseline' AD biomarker level). AD biomarkers of interest include Amyloid-Beta 1-42 (Aβ42), t-tau, and P-tau181. Should participants not have this data available at baseline, the research team will conduct a blood draw for AD biomarker levels at baseline and at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60 years or older
* Diagnosis of Mild Cognitive Impairment (MCI)
* Pittsburgh Sleep Quality Index total score >5 or Epworth Sleepiness Scale score of ≥ 10
* Read and understand English
* Have Internet and email access

Exclusion Criteria:

* No telephone access
* Must not be taking any medication known to affect rapid eye movement (REM) sleep (or sleep architecture in general)
* Use of choline supplements.
* Epilepsy or head trauma resulting in unconsciousness in the past two years
* Known allergic reactions to components of Citicoline
* Presence of chronic obstructive pulmonary disease, asthma, severe cardiac insufficiency (congestive heart failure, myocardial infarction), type I diabetes, vitamin B12 or folic acid deficiency, liver cirrhosis, thyroid dysfunction, rheumatoid arthritis, chronic renal failure, severe/unstable psychiatric disorders, moderate to severe obstructive sleep apnea, restless legs syndrome or periodic limb movement disorder
* History of alcohol dependence and drug abuse
* Night shift workers or those in situations where they regularly experience jet lag or have irregular work schedules

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Pittsburgh Sleep Quality Index (PSQI) | Baseline and 3 months
  This questionnaire is used to measure subjective sleep quality. It has strong validity and reliability in clinical populations and consists of 19 items asking about sleep disturbances over the past month with 7 dimensions. Each dimension scores 0 (no difficulty) to 3 (severe difficulty) and the sum of these scores yields a global sleep quality score that ranges from 0-21. Higher scores indicate greater difficulty sleeping. This questionnaire can be filled out by the participant, caregiver, or both as appropriate.
Change in the Epworth Sleepiness Scale (ESS) | Baseline and 3 months
  The ESS is a clinical and research standard used to assess perceived daytime sleepiness over the past month. It is a self-administered validated questionnaire and takes 2-3 minutes to fill out. Respondents are asked to rate how likely they are to doze off in 8 situations, from 0 (would never dose) to 3 (high chance of dozing). Any score of 10 or above is considered an indicator of pathologic sleepiness. This questionnaire can be filled out by the participant, caregiver, or both as appropriate.
Change in percentage of the rapid eye movement (REM) sleep | Baseline and 3 months
  The change in % REM sleep will be measured using The Sleep Profiler using the polysomnography 2 (PSG2), which is an Electroencephalogram (EEG) Sleep Monitor that is an FDA-cleared, easily applied, wireless EEG device developed and validated to measure sleep architecture for in-home sleep studies. This will be worn for 2 nights at baseline and again for 2 nights at follow-up.
Change in sleep duration | Baseline and 3 months
  Average sleep duration (hours) will be measured via a subjective 7-day sleep diary that collects subjective sleep/wake patterns and naps. It is the "gold standard" for subjective sleep assessment of sleep duration. It will be filled out by the participant in conjunction with the caregiver.
Change in plasma choline levels | Baseline and 3 months
  Blood draws will be made at baseline and follow-up.
Change in beta-amyloid 42 levels | Baseline and 3 months
  Levels of beta-amyloid 42. A lumbar puncture (LP) will be performed at 3 months in participants who have already had a previous LP. For those who don't have a previous LP performed, blood samples will be drawn before starting the study medication and at follow-up.
Change in tau and phospho-tau levels | Baseline and 3 months
  Levels of tau, and phospho-tau will be measured. A lumbar puncture (LP) will be performed at 3 months in participants who have already had a previous LP. For those who don't have a previous LP performed, blood samples will be drawn before starting the study medication and at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Pak, PhD, MS, MTR, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University School of Nursing, Atlanta, Georgia
  - Goizueta Alzheimer's Disease Research Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The research team will share deidentified data in accordance with the NIH Data Sharing Policy to share research resources (biological samples and finalized data). Deidentified data and deidentified biological samples will be stored and shared with other institutions or companies as approved by a Scientific Review Committee and in accordance with all applicable regulations.
Time Frame: Anticipated data availability will be at the conclusion of this study on 7/1/25.
Access Criteria: Data will be shared with the Aging Research Biobank. The data generated in this study will be housed in the Aging Research Biobank. The database can be found at the following link: agingresearchbiobank.nia.nih.gov
URL: https://agingresearchbiobank.nia.nih.gov

DOCUMENTS (1):
  • Informed Consent Form (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT06029894/ICF_000.pdf